CLINICAL TRIAL: NCT07326150
Title: Construction of a Predictive Model for the Efficacy of Chemoprevention Combined With Targeted Therapy in Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2025-1714（IIT）
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer Resectable; Pancreatic Cancer Non-resectable
Keywords: Chemotherapy combined with immunotherapy; efficacy prediction; Organoids; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Patient tumor tissue sections, blood and fresh tumor tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pancreatic ductal adenocarcinoma: Pancreatic cancer confirmed by pathology and imaging studies
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — 1. Blood Sample Collection: Prior to initial treatment, collect one tube of clotting blood (10 ml, serum separator tube) from the patient.
  2. Fresh Tumor Tissue: With informed consent obtained, collect pancreatic cancer or liver metastatic tissue specimens (one 2cm³ surgical specimen or one ≥1cm biopsy specimen) via surgery or biopsy prior to treatment.
  3. Tumor Tissue Sections: Retrospectively collected from our hospital's pathology department, 60 pancreatic cancer patient samples archived over the past 5 years were retrieved.

SUMMARY:
This study is a single-center, observational clinical trial designed to enroll a total of 70 pancreatic cancer patients. Tumor tissue sections from 60 patients will be retrospectively collected to establish a treatment response prediction model using spatial transcriptomics and other analyses. Fresh tumor tissue and blood samples from 10 patients will be prospectively collected to establish pancreatic cancer organoids and humanized immunocompetent mouse models for functional validation and exploration of the underlying molecular mechanisms.

DETAILED DESCRIPTION:
Primary Objective: Based on a cohort of pancreatic cancer patients receiving combined chemotherapy with immunotherapy and targeted therapy, analyze tumor microenvironment characteristics through multiplex immunohistochemistry and spatial transcriptomics. Identify key biomarkers associated with treatment efficacy and prognosis, and establish a clinically applicable predictive model for treatment outcomes in pancreatic cancer patients undergoing combined chemotherapy with immunotherapy and targeted therapy.

Secondary Objectives: Establish pancreatic cancer organoids and humanized immunocompetent mouse models to functionally validate the aforementioned efficacy prediction model and explore the molecular mechanisms by which the tumor microenvironment modulates treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pathologically and radiologically confirmed pancreatic cancer

Exclusion Criteria:

* Active malignancy other than pancreatic malignancy within the past 5 years or concurrently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer confirmed by pathology and imaging studies
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Best Tumor Response | 12 months
  Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Overall Survival | 60 months
  Overall survival is the duration from diagnosis to death. For patients who are alive, overall survival is censored at the last contact.

SECONDARY OUTCOMES:
Progression-free Survival | 36 months
  The period from diagnosis until disease progression or death on study, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
We currently have no plans to share individual participant data (IPD) with other researchers.